CLINICAL TRIAL: NCT06887842
Title: Posterior Nasal Nerve Surgical Resection Versus Radiofrequency Ablation Versus Surface Coblation for Treatment of Intractable Allergic Rhinitis
Brief Title: Posterior Nasal Nerve Neurectomy for Treatment of Intractable Allergic Rhinitis
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Ahmed Magdi Noaman Othman Orabi, Principal Investigator, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: KFSIRB200-543
Record Dates: First submitted 2025-03-09; First posted 2025-03-20 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-03

CONDITIONS: Intractable Allergic Rhinitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Posterior nasal neurectomy by surgical resection (Active Comparator)
  Interventions: Device: Posterior Nasal Nerve neurectomy
- Posterior nasal neurectomy by radio- frequency ablation (Active Comparator)
  Interventions: Device: Posterior Nasal Nerve neurectomy
- Surface coblation on area of the course of the Posterior nasal nerve (Active Comparator)
  Interventions: Device: Posterior Nasal Nerve neurectomy

INTERVENTIONS:
Device: Posterior Nasal Nerve neurectomy — Posterior Nasal Nerve neurectomy which is done by surgical resection.
  Arms: Posterior nasal neurectomy by surgical resection
Device: Posterior Nasal Nerve neurectomy — Posterior Nasal Nerve neurectomy which is done by using radiofrequency ablaion.
  Arms: Posterior nasal neurectomy by radio- frequency ablation
Device: Posterior Nasal Nerve neurectomy — Posterior Nasal Nerve neurectomy by coblation of the surface of the course of the nerve
  Arms: Surface coblation on area of the course of the Posterior nasal nerve

SUMMARY:
This study aims to compare the outcomes of posterior nasal nerve neurectomy in patients with resistant Allergic rhinitis by using three different methods ( surgical resection vs radiofrequency ablation vs surface coblation ) through assesment of functional outcomes, postoperative complications, and impacts on quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 16 to 65 years, fit for surgery, diagnosed as moderate to severe persistent Allergic Rhinitis, as per the ARIA guidelines having 3 or more of the typical symptoms of Allergic Rhinitis including nasal discharge, repeated attacks of sneezing, nasal itching and nasal obstruction.

Exclusion Criteria:

* • Patients with Coexisting nasal pathologies that could influence the outcomes of the surgery like: chronic granulomatous diseases of the nose, nasal tumors, chronic sinsitis with or without nasal polyps, etc.

  * Patients who had used topical steroid nasal spray, oral or topical antihistamines, oral leukotriene antagonists, oral or tobical nasal decongestants in the last 2 weeks.
  * Immunocompromised patients, Systemic disease affecting prognosis such as diabetes mellitus, hypertension,chronic liver failure or heart failure.
  * Unwillingness for endoscopic surgery.
  * Patients younger than 18 years of age.
  * Patients who are unfit for general anesthesia.
  * Previous history of nasal surgery

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-04-25 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Improvement of the four main symptoms (Sneezing ,itching , rhinorrhea ,nasal obstruction) | Evaluations will be scheduled for 2 weeks, one month, three months, and six months following surgery.
  These symptoms will be assessed using the SNOT-22 rhinologic subdomain questionnaire which is routinely and prospectively administered to all patients, and individual item scores within the rhinologic subdomain (need to blow nose, sneezing, runny nose, cough, post- nasal discharge, and thick nasal discharge) will be tabulated, each symptom will be scored on a scale from 0 to 5 (0 = no problem, 1 = very mild problem, 2 = mild problem, 3 = moderate problem, 4 = severe problem and 5 = problem as bad as it can be).

SECONDARY OUTCOMES:
postoperative complications eg. Bleeding, crustations etc, postoperative endoscopic score will be evaluated. | 2 weeks, 1M month after the procedure .
  Bleeding assessment using The Modena bleeding score. Postoperative endoscopic score including : (discharge, crust formation ,scarring ) after the operation will be also recorded and documented using the LundKennedy (LK) system.

CONTACTS AND LOCATIONS:
Locations (1):
- kafrelsheikh University Hospitals, Kafrelsheikh, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ahilasamy N, Rajendran Dinesh K. [Endoscopic posterior nasal neurectomy]. J Laryngol Otol. 2019 Sep;133(9):825-829. doi: 10.1017/S002221511900166X. Epub 2019 Aug 23. Spanish. PMID 31439065